CLINICAL TRIAL: NCT04326374
Title: The Efficacy, Safety and Tolerability of TransCon hGH Administered Weekly Versus Daily hGH in Prepubertal Children With Growth Hormone Deficiency: a Randomized, Open-lable, Active-controlled, Parallel-group Study in China
Brief Title: Safety, Tolerability and Efficacy of TransCon hGH Weekly Versus Daily hGH in Chinese Pediatric Growth Hormone Deficiency
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Visen Pharmaceuticals (Shanghai) Co., Ltd. (Industry)
Collaborators: Ascendis Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT301-CN; CTR20200399 (Other: Center for drug evaluation,NMPA)
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Growth Hormone Deficiency; Endocrine System Diseases; Hormones; Pituitary Diseases; Pituitary Disease, Anterior
Keywords: Growth Hormone Deficiency; TransCon hGH; human growth hormone; hGH
MeSH Terms: conditions — Dwarfism, Pituitary; Endocrine System Diseases; Pituitary Diseases | interventions — lonapegsomatropin; Human Growth Hormone; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be randomized to 1 of the 2 treatment groups: either weekly TransCon hGH or daily hGH, in a 2:1 ratio
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TransCon hGH (Experimental): TransCon hGH will be self-administered or injected by parents once weekly. The dose will be adjusted based on subject's weight.
  The treatment will continue 52 weeks.
  Interventions: Drug: TransCon hGH
- Daily hGH (Active Comparator): Daily hGH will be self-administered or injected by parents once daily. The dose will be adjusted based on subject's weight.
  The treatment will continue 52 weeks.
  Interventions: Drug: daily hGH

INTERVENTIONS:
Drug: TransCon hGH — Once weekly subcutaneous injection
  Other Names: ACP-011
  Arms: TransCon hGH
Drug: daily hGH — Once daily subcutaneous injection
  Other Names: somatropin (rDNA orgin) for injection
  Arms: Daily hGH

SUMMARY:
This study is conducted in China only. The purpose is to demonstrate the efficacy and safety of once weekly dosing of TransCon hGH, a long-acting growth hormone product, compare to once-daily dosing of human growth hormone (hGH) after 52 weeks of treatment in prepubertal children with growth hormone deficiency (GHD).

DETAILED DESCRIPTION:
Not Provided

ELIGIBILITY:
Inclusion Criteria:

* Prepubertal children with GHD in Tanner stage 1, aged of 3 years and below 17 years;
* Impaired HT defined as at least 2.0 standard deviations (SD) below the mean height for chronological age and sex (HT SDS≤-2.0) according to the Chinese 2005 standard；
* Diagnosis of GHD confirmed by 2 different GH stimulation tests, defined as a peak GH level of ≤10 ng/mL, determined with a validated assay. Bone age (BA) at least 6 months less than the chronological age；
* Baseline IGF-1 level of at least 1.0 SD below the mean IGF-1 level standardized for age and sex (IGF-1 SDS ≤-1.0)；
* Written, signed informed consent of the parent(s) or legal guardian(s) of the subject and written assent of the subject (if the subject is 8 years old or above).

Exclusion Criteria:

* Children with a body weight below 12 kg；
* Prior exposure to recombinant hGH or IGF-1 therapy；
* Children with past or present intracranial tumor growth as confirmed by a sellar MRI scan (with contrast dye recommended) at Screening
* Children born SGA (birth weight ≤10th percentile for gestational age according to the Chinese reference)；
* Children with psychosocial dwarfism；
* Children with idiopathic short stature；
* Other causes of short stature such as coeliac disease, hypothyroidism, or rickets；
* History or presence of malignant disease; any evidence of present tumor growth;
* Subjects with diabetes mellitus；
* Closed epiphyses；
* Major medical conditions and/or presence of contraindication to hGH treatment；
* Participation in any other trial of an investigational agent within 3 months prior to Screening.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2019-12-30 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Annualized height velocity(AHV) at Week 52 | 52 Weeks
  Annualized height velocity at Week 52 for weekly TransCon hGH treatment and the daily hGH treatment groups

SECONDARY OUTCOMES:
AHV and the change from baseline over 52 weeks at each visit | 52 Weeks
  AHV and the change from baseline for the TransCon hGH and the daily hGH treatment group over 52 weeks at each visit
Height SDS and the change from baseline over 52 weeks | 52 weeks
  Height SDS and the change from baseline for the TransCon hGH and the daily hGH treatment group over 52 weeks
Serum IGF-1 and IGFBP-3 levels, and IGF-1 SDS, IGFBP-3 SDS, and the change from baseline over 52 weeks at each visit | 52 weeks
  Serum IGF-1 and IGFBP-3 levels, and IGF-1 SDS, IGFBP-3 SDS, and the change from baseline for the TransCon hGH and the daily hGH treatment group over 52 weeks at each visit
The percentage of participants achieving IGF-1 SDS 0 to +2.0 | 52 weeks
  The normalization of IGF-1 SDS (percentage of participants achieving IGF-1 SDS 0 to +2.0 over 52 weeks for the TransCon hGH and the daily hGH treatment group
Incidence of Treatment-Emergent Adverse Events | 52 weeks
The plasma concentration | 52 weeks
  pharmacokinetics measure of hGH over 52 weeks in TransCon hGH group

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Luo, MD, Principal Investigator — Tongji Hospital
Locations (1):
- Department of Pediatrics, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology,, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No